CLINICAL TRIAL: NCT03161912
Title: An Observational Study Program to Investigate the Effectiveness of Intravitreal Aflibercept in Diabetic Macular Edema and/or Macular Edema Secondary to Retinal Vein Occlusion in a Real World Setting
Brief Title: A Study to Evaluate the Effectiveness of Intravitreal Aflibercept in Patients With Diabetic Macular Edema and/or Macular Edema Secondary to Retinal Vein Occlusion, Which Either Have or Have Not Been Pretreated for Their Disease
Acronym: AURIGA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 19157
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Macular Edema
Keywords: Diabetes; Retinal Diseases; Diabetic Retinopathy; Diabetic macular edema; Retinal vein occlusion; Macular edema secondary to retinal vein occlusion; Intravitreal anti-VEGF (vascular endothelial growth factor); VEGF inhibitor; aflibercept; real world data; treatment pattern
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus; Retinal Diseases; Diabetic Retinopathy; Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DME/naïve: patients with pre-treatment in diabetic macular edema (DME)
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- DME/pre-treatment: patients without pre-treatment in DME
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- RVO/pre-treatment: Macular edema secondary to RVO with prior treatment
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- RVO/naïve: Macular edema secondary to RVO without prior treatment
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — As per the treating physicians discretion.

SUMMARY:
AURIGA is designed to collect data from routine clinical practice on the effectiveness and utilization of intravitreal aflibercept in the treatment of visual impairment due to diabetic macular edema (DME) or macula edema secondary to retinal vein occlusion (RVO).

The primary objective of this observational study (OS) is to evaluate the effectiveness of intravitreal aflibercept in 4 cohorts (with/without prior treatment in DME or macular edema secondary to RVO) in each of the participating countries.

Additionally, utilization and treatment regimens in routine clinical practice will be described.

Health care resources and services as well as health out-comes related to vision loss will be evaluated based on information collected using the AURIGA patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* For DME

  -- Female and male patients of legal age, as defined by local regulations and local product labels, with visual impairment due to DME
* For macular edema secondary to RVO

  -- Female and male patients of legal age, as defined by local regulations and local product labels, with visual impairment due to macular edema secondary to RVO
* Patient for whom the decision to initiate treatment with aflibercept is made prior to and independent from study participation
* Signed informed consent.

Exclusion Criteria:

* Any contraindications as listed in the local intravitreal aflibercept SmPC (summary of product characteristics)
* Current participation in any other clinical (interventional) study or in any other anti-VEGF study
* Receipt of systemic anti-VEGF and pro-VEGF treatment
* Structural damage to the center of the macula in either eye that is likely to preclude improvement in VA following the resolution of macular edema or any other condition expected to permanently limit VA outcomes over the course of the study
* Patients with prior retinal surgery
* Any prior treatment with aflibercept
* History of stroke or transient ischemic attacks within the last 6 months
* Laser photocoagulation (panretinal or macular) in the study eye within 90 days of Day 1
* For patients with prior treatment (i.e. patients that previously have been treated with intravitreal anti-VEGF or steroids):

  * Previous treatment of the study eye with anti-angiogenic drugs or laser within the last 3 months and patients with ocular surgery of the study eye within the last 3 months
  * Intravitreal dexamethasone or triamcinolone in the study eye within the last 3 months
  * Fluocinolone implant within the last 3 years
  * Dexamethasone implant within the last 6 months
* For DME

  -- Concomitant therapy with any other agent to treat DME in the study eye.
* For macular edema secondary to RVO

  * Patients who have received or who require pan retinal photocoagulation due to neovascularization
  * Concomitant therapy with any other agent to treat macular edema secondary to RVO in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients of legal age with a diagnosis of DME or macular edema following RVO will be enrolled in eye clinics and ophthalmology practices after the decision for treatment with aflibercept has been made by the treating physician.
Sampling Method: Probability Sample
Enrollment: 2481 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity (VA) from baseline to 12 months as evaluated in routine clinical practice per cohort and per country. | Baseline and at 12 months
  Analysis will be done per cohort and country.

SECONDARY OUTCOMES:
Mean change of visual acuity from baseline to 6, 12 and 24 months after first treatment | Up to 24 months
  Secondary endpoint based on a pooled analysis over all countries and cohorts.
Percentage of study eyes with pre-determined VA gains and losses (equivalent to 5, 10 and 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters closest to the visit 6, 12 and 24 months after first treatment | Up to 24 months
  Analysis will be done per cohort and country.
Mean change from baseline in central retinal thickness (CRT) as measured with optical coherence tomography (OCT) to closest to the visit 6, 12 and 24 months after first treatment | Up to 24 months
  Analysis will be done per cohort and country.
Proportion of study eyes with no fluid persistence as measured by spectral domain OCT (SD-OCT) closest to the visit 6, 12, and 24 months after first treatment | Up to 24 months
  Analysis will be done per cohort and country.
Treatment pattern based on the number of intravitreal aflibercept injections in the study eye during the first 6 months, the first year, and the 2-year treatment period | Up to 2 years
  Analysis will be done per cohort and country.
Mean number of visits regarding the study eye by type of visit during the first 6 months, the first year, and the 2-year treatment period | Up to 2 years
  Analysis will be done per cohort and country. Including number of visits in clinics/ophthalmology practices other than the study center.
Number of visits regarding the study eye in clinics/ophthalmology practices other than the study center during the first 6 months, the first year, and the 2-year treatment period | Up to 2 years
Number of procedures per patient during the first 6 months, the first year, and the 2-year treatment period | Up to 2 years
  Analysis will be done per cohort and country.
  The procedures contains:
  * Slit lamp biomicroscopy
  * Funduscopy examination
  * Fluorescein angiographies
Number of patients requiring additional drug treatment and what category of drug (patients switching to steroid treatment only or to other anti-VEGFs are excluded) | Up to 2 years
  Analysis will be done per cohort and country.
Number of performed laser treatments | Up to 2 years
  Analysis will be done per cohort and country.
Treatment pattern based on mean time between visits and mean time between aflibercept injections | Up to 2 years
  Analysis will be done per cohort and country.
Mean change in VA by number of injections during the first 6 months, the first year, and the 2-year treatment period. | Up to 2 years
  Analysis will be done per cohort and country.

CONTACTS AND LOCATIONS:
Locations (11):
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Egypt
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Kuwait
- Many Locations, Multiple Locations, Lebanon
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Saudi Arabia
- Many Locations, Multiple Locations, Taiwan
- Many Locations, Multiple Locations, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Donati S, Yang CH, Xu X, Mura M, Giocanti-Auregan A, Hoerauf H, Allmeier H, Machewitz T, Johnson KT, Santoro E; AURIGA study investigators. Intravitreal Aflibercept for the Treatment of Diabetic Macular Edema in Routine Clinical Practice: Results from the 24-Month AURIGA Observational Study. Ophthalmol Ther. 2024 Jan;13(1):161-178. doi: 10.1007/s40123-023-00829-3. Epub 2023 Nov 4. PMID 37924483
- [Derived] Giocanti-Auregan A, Donati S, Hoerauf H, Allmeier H, Rittenhouse KD, Machewitz T, Yang CH; AURIGA Study Investigators. Real-World Management of Macular Edema Secondary to Retinal Vein Occlusion with Intravitreal Aflibercept: 24-month Results from the AURIGA Observational Study. Ophthalmol Ther. 2024 Jan;13(1):179-203. doi: 10.1007/s40123-023-00830-w. Epub 2023 Nov 4. PMID 37924481